CLINICAL TRIAL: NCT00213915
Title: Effects of Oral Chronic L-arginine Supplementation on Exercise and Renal Function of Heart Transplant Recipients
Brief Title: L-arginine Supplementation and Exercise; L-arginine Supplementation and Renal Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3031
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Heart Transplantation
Keywords: L-arginine; exercise capacity; renal function; nitric oxide; exercise capacity using a maximal exercise test; urinary elimination of a saline load using blood and urinary samples

INTERVENTIONS:
Drug: 12 g of L-arginine glutamate during 6 weeks twice a day

SUMMARY:
* exercise capacities are still altered after heart transplantation partly due to peripheral endothelial dysfunction
* cyclosporin-induced renal dysfunction may be due to renal endothelial dysfunction and can be reversed in an animal model by L-arginine supplementation
* to determine the potential beneficial effect of L-arginine supplementation on exercise capacity and renal function of heart transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Male (> 18 years old) stable heart transplant recipient for at least 6 weeks
* Stable treatment for at least 3 months
* Sedentary people

Exclusion Criteria:

* Unstable cardiac pathology
* Obesity (IMC > 40)
* Participation in another study in the last month
* Chronic renal failure (creatinine clearance < 20 ml/min)
* Renal transplantation
* Diabetes
* Impossibility to practice exercise test
* Nitrate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-02 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Maximal and sub maximal exercise capacity at the end of the 6 weeks L-arginine supplementation. Renal function at the end of the 6 weeks

SECONDARY OUTCOMES:
No secondary effects

CONTACTS AND LOCATIONS:
Overall Officials: Stephane DOUTRELEAU, MD, Principal Investigator — Service de Physiologie et d'Explorations Fonctionnelles
Locations (3):
- France (3):
  - Institut de Physiologie, Strasbourg
  - Service de Chirurgie Vasculaire, Strasbourg
  - Service des Explorations Fonctionnelles Respiratoires et de l'Exercice, Strasbourg

REFERENCES:
- [Result] Doutreleau S, Rouyer O, Di Marco P, Lonsdorfer E, Richard R, Piquard F, Geny B. L-arginine supplementation improves exercise capacity after a heart transplant. Am J Clin Nutr. 2010 May;91(5):1261-7. doi: 10.3945/ajcn.2009.27881. Epub 2010 Mar 3. PMID 20200265